CLINICAL TRIAL: NCT06486623
Title: Effect of Supplementation With Anthocyanins Contained in Black Chokeberry (Aronia Melanocarpa) on Selected Indicators of Iron Metabolism in Female Swimmers
Brief Title: Effect of Supplementation With Anthocyanins on Iron Metabolism in Female Swimmers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: MMydłowska_PhD
Record Dates: First submitted 2024-02-06; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-01

CONDITIONS: Iron Deficiencies; Inflammation; Oxidative Stress; Female Athlete Triad
MeSH Terms: conditions — Iron Deficiencies; Inflammation; Female Athlete Triad Syndrome | interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Supplemented group (Experimental): The supplemented group (n=12) consumed capsules with highly concentrated 18% chokeberry extract (one capsule contained 200 mg). Each capsule also contained: chokeberry fiber, E460b magnesium salts of stearic acid (anti-caking agent), E551 silicon dioxide (anti-caking agent), hydrocypropyl methylcellulose (capsule shell) and E171 titanium dioxide (shell colour). The producer of all capsules is MLD Biotrade in Poznan.
  The swimmers took 2 capsules a day (before breakfast and dinner) for nearly 56 days (depending on length menstrual cycle phase). The swimmers sipped each capsule with glass of water.
  Interventions: Drug: Black chokeberry extract in capsules with 18% standardization of the anthocyanins content
- 2. Placebo group (Placebo Comparator): The control group (n=10) consumed capsules that were made from chokeberry fiber. The producer of all capsules is MLD Biotrade in Poznan.
  The swimmers took 2 capsules a day (before breakfast and dinner) for nearly 56 days (depending on length menstrual cycle phase). The swimmers sipped each capsule with glass of water.
  Interventions: Drug: Chokeberry fiber in capsules

INTERVENTIONS:
Drug: Black chokeberry extract in capsules with 18% standardization of the anthocyanins content — Supplement group: supplement of diet - black chokeberry extract (capsules) with 18% standardization of the anthocyanins content (one capsule contained 200 mg). Each capsule also contained: chokeberry fiber, E460b magnesium salts of stearic acid (anti-caking agent), E551 silicon dioxide (anti-caking agent), hydrocypropyl methylcellulose (capsule shell) and E171 titanium dioxide (shell colour).
  The producer of all capsules is MLD Biotrade in Poznan.
  Other Names: Aronia melanocarpa
  Arms: 1. Supplemented group
Drug: Chokeberry fiber in capsules — Placebo group: placebo product - chokeberry fiber (placebo capsules, which were made from chokeberry fiber).
  The producer of all capsules is MLD Biotrade in Poznan.
  Other Names: Placebo product
  Arms: 2. Placebo group

SUMMARY:
The study included 8-weeks supplementation of black chokeberry extract with 18% standardization of the anthocyanins content (dose 2×200 mg per day), or a placebo product that was made from chokeberry fiber.

Purpose:

The aim of the study is effectiveness check of black chokeberry intake as a potential factor which, due to its ability to reduce inflammation and chelate iron ions, will have an impact on minimizing undesirable changes in the red blood cell system.

Hypothesis:

Main hypothesis: Supplementation of black chokeberry (Aronia melanocarpa) has a positive effect on iron economy of female swimmers.

Auxiliary hypotheses:

1. Supplementation of black chokeberry enhances the antioxidant status and has a positive effect on the prooxidant-antioxidant balance.
2. Supplementation of black chokeberry reduce inflammation induced by intensive exercises, by reducing inflammatory markers.

Study plan:

Before first term of the study:

Control of Menstrual Cycle Phases since March 2023 (installing the application on the phone - Menstrual Period Tracker calendar).

First term of the study:

1. Menstrual cycle control survey.
2. Conduct a body composition analysis.
3. Collection of blood samples before the exercise test for biochemical determinations.
4. Exercise test in the swimming pool - crawl style intensive test (800 m + 200 m + 50 m).
5. Collection of blood immediately after exercise and 3 hours later.
6. Supplementation for nearly 56 days, depending on the length of the menstrual cycle.

Second term of the study:

Repeat the measurements from the 1st date of test.

Participants: The group of selective and homogeneous female swimmers, who train swimming intensively and attend the Sports Championship School Complex.

DETAILED DESCRIPTION:
This study included 8-weeks supplementation of black chokeberry extract with 18% standardization of the anthocyanins content (dose 2×200 mg per day), or a placebo product that was made from chokeberry fiber. The first date of research completed the group of twenty-four and homogeneous female swimmers, who train swimming intensively and attend the Sports Championship School Complex. The second date of research completed the group of twenty-two selective and homogeneous female swimmers, who train swimming intensively and attend the Sports Championship School Complex.

Purpose:

The aim of the study is effectiveness check of black chokeberry intake as a potential factor which, due to its ability to reduce inflammation and chelate iron ions, will have an impact on minimizing undesirable changes in the red blood cell system.

Hypothesis:

Main hypothesis: Supplementation of black chokeberry (Aronia melanocarpa) has a positive effect on iron economy of female swimmers.

Auxiliary hypotheses:

1. Supplementation of black chokeberry enhances the antioxidant status and has a positive effect on the prooxidant-antioxidant balance.
2. Supplementation of black chokeberry reduce inflammation induced by intensive exercises, by reducing inflammatory markers.

The research is going to be carried out as a medicinal experiment with tissue interference (approval of Research Ethics Committee: 538/22 of 06/23/2022, with changes: 221/23 of 03/09/2023). All swimmers qualified to study based on inclusion and exclusion criteria and were informed of the extract course of the study and gave written consent to participate.

EXPERIMENTAL PROCEDURE, WHICH WAS APPLIED (STUDY PLAN):

A. Before first term of the study:

Control of Menstrual Cycle Phases since March 2023 (installing the application on the phone - Menstrual Period Tracker calendar) and three surveys in three terms.

B. First term of the study:

1. Menstrual cycle control by application Menstrual Tracker Period Calendar and surveys, before swimming test.
2. Body composition analysis (TANITA MC-780 S MA).
3. Biochemical determinations - blood samples will be taken before and after exercise test as well as after 3-hour restitution, in order to determine:

   * morphological parameters,
   * value of indicators:

     1. iron status problems (iron, hepcidin, erythroferrone, total iron-binding capacity, unsaturated iron-binding capacity, ferritin, transferrin,
     2. oxidative stress (total antioxidant capacity),
     3. immunological indicators (interleukins: IL-6, IL-2, IL-10, C-reactive protein),
     4. hormonal balance (progesterone, estradiol, luteinizing hormone, follicle-stimulating hormone),
     5. other: lactic acid, myoglobin, hypoxanthine.

   Blood samples were collected from the elbow vein into two 4-ml tubes (to obtain serum) and centrifuged at 3,000 rpn and into 2,7-ml tubes to determine morphology. Morphology was determined on the same day the samples were collected, while serum was frozen and stored at -80 Celsius degrees until assays were performed. In addition, before and immediately after the exercise test, capillary blood was drawn from the earlobe to determine lactate levels.

   Lactate level were determined immediately after capillary blood sampling using a commercial available kit (Dr Lange, Germany). The concentration of lactate was determined in mmol/l. Other measurements were determined using ELISA kits (DRG Medtek).
4. Intensive exercise test in the swimming pool, before supplementation - crawl style (800 m + 200 m + 50 m) with 15-minute active rest between test sections.
5. Supplementation of black chokeberry - nearly 56-days supplementation of black chokeberry extract with 18% standardization of the anthocyanins content (connection with menstrual cycle phase).The swimmers were randomly divided into two groups: supplementation and placebo. The placebo contained chokeberry fiber. Whole products were manufactured by MLB BIOTRADE, Poznan. The swimmers took 2 capsules per day (before breakfast and dinner) and they sipped each capsule with glass of water.

C. Second term of the study:

1. Menstrual cycle control by application Menstrual Tracker Period Calendar and surveys, before swimming test.
2. Body composition analysis (TANITA MC-780 S MA).
3. Biochemical determinations - blood samples will be taken before and after exercise test as well as after 3-hour restitution, in order to determine:

   * morphological parameters (erythrocytes, leukocytes, thrombocytes),
   * value of indicators responsible for:

     1. iron status problems (iron, hepcidin, erythroferrone, total iron-binding capacity, unsaturated iron-binding capacity, ferritin, transferrin),
     2. oxidative stress (total antioxidant capacity),
     3. immunological indicators (interleukins: IL-6, IL-2, IL-10, C-reactive protein (CRP)),
     4. hormonal balance (progesterone, estradiol, luteinizing hormone (LH), follicle-stimulating hormone (FSH)),
     5. other: lactic acid, myoglobin, hypoxanthine.

   Blood samples were collected from the elbow vein into two 4-ml tubes (to obtain serum) and centrifuged at 3,000 rpn and into 2,7-ml tubes to determine morphology. Morphology wa determined on the same day the samples were collected, while serum was frozen and stored at -80 Celsius degrees until assays were performed. In addition, before and immediately after the exercise test, capillary blood was drawn from the earlobe to determine lactate levels.

   Lactate level were determined immediately after capillary blood sampling using a commercial available kit (Dr Lange, Germany). The concentration of lactate was determined in mmol/l. Other measurements were determined using ELISA kits (DRG Medtek).
4. Intensive exercise test in the swimming pool, after supplementation - crawl style (800 m + 200 m + 50 m) with 15-minute active rest between test sections.

Data collection, analysis in laboratory, statistical analysis and preparation articles to publication.

ELIGIBILITY:
Inclusion Criteria:

* Current medical examinations issued by a sports medicine doctor
* Training experience a minimum of three years
* Student of a sports championship school team
* Consent of the athlete/legal guardian to participate in the research
* Completion of the exercise test in the swimming pool - crawl style intensive test (800 m + 200 m + 50 m) on two test deadline

Exclusion Criteria:

* Taking: oral contraceptive pills, supplements containing anthocyanin compounds during the study or a one month earlier
* Health problems
* Antibiotic therapy

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Physiological parameters of blood morphology I | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  erythrocytes: RBC [10^6/mL], HGB [g/dL], HCT [%], MCV [mm^3], MCH [pg], MCHC [g/dL], RDW [%],
Physiological parameters of blood morphology II | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  leukocytes: WBC [10^3/mL], LYM [10^3/mL], MON [10^3/mL], GRA [10^3/mL], LYM [%], MON [%], GRA [%],
Physiological parameters of blood morphology III | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  thrombocytes: PLT [10^3/mL], MPV [mm^3], PCT [%], PDW [%]
Physiological parameters of iron metabolism indicator I | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  iron [µg/dl]
Physiological parameters of iron metabolism indicator II | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  hepcidin [ng/ml]
Physiological parameters of iron metabolism indicator III | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  transferrin [mg/ml]
Physiological parameters of iron metabolism indicator IV | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  total iron-binding capacity (TIBC) [µg/dl]
Physiological parameters of iron metabolism indicator V | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  ferritin [ng/ml]
Physiological parameters of iron metabolism indicator VI | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  erythroferrone [ng/mL]
Physiological parameters of antioxidant-prooxidant indicator | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  total antioxidant capacity [mmol/l]
Physiological parameters of immunological indicator I | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  interleukin 6 [ng/L]
Physiological parameters of immunological indicator II | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  interleukin 2 [ng/L]
Physiological parameters of immunological indicator III | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  interleukin 10 [ng/L]
Physiological parameters of immunological indicator IV | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  C-reactive protein [mg/dL]
Physiological parameter of hormonal indicator I | At each exercise test (up to 15 minute before exercise)
  progesterone [ng/ml]
Physiological parameter of hormonal indicator II | At each exercise test (up to 15 minute before exercise)
  estradiol [pg/ml]
Physiological parameter of hormonal indicator III | At each exercise test (up to 15 minute before exercise)
  luteinizing hormone (LH) [mIU/ml]
Physiological parameter of hormonal indicator IV | At each exercise test (up to 15 minute before exercise)
  follicle-stimulating hormone (FSH) [mIU/ml]
Other physiological parameter I | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  myoglobin [ng/ml]
Other physiological parameter II | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  hypoxanthine [mmol/l]
Other physiological parameter (with capillary blood - earlobe) | At each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  lactic acid [mmol/l]

SECONDARY OUTCOMES:
Physiological parameters of iron metabolism indicator VII | Calculated with blood samples at each exercise test (up to 15 minute before exercise, up to 1 minute post exercise, 3 hours after)
  unsaturated iron-binding capacity (UIBC)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Mydłowska, PhD student, Principal Investigator — Poznań University of Physical Education, Faculty of sport sciences in Gorzów Wielkopolski
Locations (1):
- University of Physical Education in Poznan, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No